CLINICAL TRIAL: NCT01948544
Title: A Study to Evaluate Improvement in the Quality of Life and Outcomes of Patients Diagnosed With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Portable Oxygen Concentrator to Improve Quality of Life in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: StratiHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: 01053013A
Record Dates: First submitted 2013-07-19; First posted 2013-09-23 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: COPD
Keywords: COPD; LTOT; Long-Term Oxygen Therapy; Portable Oxygen Concentrator; Quality of Life; Six Minute Walk Distance Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic obstructive pulmonary disease: * More than 12 million adults are diagnosed with COPD
  * COPD is the 4th leading cause of death in the U.S.
  * Breathing difficulty is the major reason patients seek medical attention
  * COPD patients requiring hospitalization were associated with higher costs
  * Oximetry is an important tool for assessing need for Long-term oxygen therapy
  * LTOT has been proven to improve survival and quality of life
  * Patients will be provided a lightweight portable oxygen concentrator to:
    1. support increased activity
    2. improve quality of life
    3. increase functional capacity

SUMMARY:
* Evaluate subjects in an prospective observational study
* Subjects will be administered scientifically validated questionnaires
* Determine the affect of the Portable Oxygen Concentrator (POC) on improvements in:

  1. Exercise capability, dyspnea and quality of life as primary endpoints
  2. Utilize:

     1. Baseline Dyspnea Index (BDI)
     2. Transitional Dyspnea Index (TDI)
     3. Chronic Respiratory Disease Questionnaire (CRQ)
     4. Six minute walk test (6MWT)
     5. Epworth Sleepiness Scale (ESS)
* The secondary endpoints will be:

  1. Rate of exacerbations, sleep quality
  2. Health care utilization (emergency room encounters, hospital admissions)

DETAILED DESCRIPTION:
Evaluate subjects in an prospective observational study in which subjects will be screened and administered scientifically validated questionnaires at study entry and during the observation period at specified intervals to determine the affect of the Portable Oxygen Concentrator on improvements in exercise capability, dyspnea and quality of life as primary endpoints, utilizing the Baseline Dyspnea Index (BDI), Transitional Dyspnea Index (TDI), the Chronic Respiratory Disease Questionnaire (CRQ) and six minute walk test (6MWT). The secondary endpoints will be rate of exacerbations, sleep quality (reported as number of hours sleep improvement; utilize Epworth Sleepiness Scale [ESS]), and health care utilization (emergency room encounters, hospital admissions).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of chronic obstructive pulmonary disease (COPD)
* Clinically stable disease at the time of consent
* Current prescription of oxygen; with previous or current oximetry suggesting desaturation at rest or during exercises (oxygen saturation ≤88% on at least one occasion)
* Highest measured FEV1, 70% predicted; and
* Highest measured FEV1/FVC, 70% predicted
* Capable of giving informed consent
* Currently using oxygen system that is either a portable tank; liquid or other Portable Oxygen Concentrator (POC)
* Mobility without a walker, cane or rollator
* Spo2 ≥ 92% on Portable Oxygen Concentrator (POC) at rest and activity
* Non-smoker at time of consent

Exclusion Criteria:

* Cardiovascular disease as defined in New York Heart Association Functional Class III
* Degenerative bone or joint disease that limits mobility and ability to perform activities of daily living and/or exercise
* Current homeless persons
* Active drug/alcohol dependence
* Recent abuse history within the past two years
* Clinically unstable at the time of consent
* Currently a tobacco smoker

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: COPD Patients prescreened and selected by their primary care physician or pulmonologist
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 6 months
  Change in functional capability, dyspnea - BDI/TDI
  • Change in exercise capability - 6MWT
Quality of Life Using Chronic Respiratory Disease Questionnaire | Measure Dyspnea at baseline upon study entry and change from baseline every two weeks up to three months; Numerical, 7-point modified Likert Scale; Total score and subscores on categories; higher scores indicate better health-related quality of life
  Quality of life - Chronic Respiratory Disease Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Pereira, MD, Principal Investigator — Tri-City Medical Center
Locations (3):
- United States (3):
  - Tri-City Pulmonary Medical Group, Oceanside, California
  - Cardinal Medical Group, Vista, California
  - Pathway Medical Group, Westminster, California